CLINICAL TRIAL: NCT06457113
Title: Augmentation of Emotional Attention Bias Modification With Targeted Memory Reactivation for Alcohol Use Disorder (AUD)
Brief Title: Emotional Attention Bias Modification and Targeted Memory Reactivation in Alcohol Use Disorder
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MZhao-018
Record Dates: First submitted 2024-06-08; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-06

CONDITIONS: Alcohol Use Disorder
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TMR group (Experimental): Patients will receive a sound S1 and sound S2 while they generate a correct outcome of Emotional Attention Bias Modification(EABM). They will also receive the sound S1 and sound S2 during REM sleep.
  Interventions: Behavioral: Emotional Attention Bias Modification and Targeted memory reactivation during REM sleep
- Control group (Active Comparator): Patients will not receive the sound S1 and sound S2 while they generate a correct outcome of Emotional Attention Bias Modification(EABM). During REM sleep, they will receive the same sound as the experimental group (S1 and S2) under the same conditions.
  Interventions: Behavioral: Emotional Attention Bias Modification

INTERVENTIONS:
Behavioral: Emotional Attention Bias Modification and Targeted memory reactivation during REM sleep — Emerging evidence shows that REM sleep is crucial for processing emotional memories and consolidating implicit memories. By using targeted memory reactivation (TMR), a known method where sound S1 and sound S2 are associated with a waking experience(i.e.negative emotional words is associated with alcohol-related cues and positive emotional words is associated with healthy lifestyle cues) and strengthened during REM sleep, the investigators aim to augment the control of craving levels in patients with Alcohol Use Disorder.
  Arms: TMR group
Behavioral: Emotional Attention Bias Modification — These patients will receive the treatment of emotional attention bias modification (EABM) without association with the sound S1 and sound S2.
  Arms: Control group

SUMMARY:
Through this protocol, researchers examine whether Targeted Memory Reactivation (TMR), a technique used to enhance memory, can augment the control of craving levels in patients with Alcohol Use Disorder by enhancing positive emotional attention bias modification.

DETAILED DESCRIPTION:
This protocol uses TMR during REM sleep to strengthen associative memories generated by emotional attention bias modification (EABM), an effective treatment for controlling craving levels in patients with Alcohol Use Disorder (AUD). EABM involves exposure to negative emotional words (e.g., frustrated, inferior) associated with alcohol-related cues and positive emotional words (e.g., successful, confident) associated with healthy lifestyle cues. The goal is to reduce alcohol-related cue positive emotional attention bias (EABs). In EABM training, alcohol-related cues and healthy activity (e.g., exercising, reading, playing musical instruments) images are always paired with negative words and positive words, respectively. The TMR group receives the EABM protocol with auditory cue feedback (sound S1-Alcohol; sound S2-Healthy Life); the control group receives the EABM protocol without auditory cue feedback. All patients will perform EABM every evening and will be exposed to sounds S1 and S2 during REM sleep with a wireless headband, which automatically detects sleep stages. Clinical evaluation of the EAB and craving levels of AUD will be conducted before and after (with a 2-week follow-up). The investigators hypothesize that patients treated with EABM and who are exposed during REM sleep to a sound that had previously been associated with the new negative memory of alcohol and the positive memory of a healthy lifestyle (TMR group) will have more reduced EAB and craving levels compared to participants exposed to the same, but non-associated, sound during REM sleep (control group).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-55 years; Meets the diagnostic criteria for Alcohol Use Disorder according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5) (American Psychiatric Association, 2013); Alcohol withdrawal period of less than 6 months; Normal vision and hearing, or corrected to normal; Agrees to participate in the study and is able to cooperate to complete the experiment.

Exclusion Criteria:

* Acute alcohol withdrawal period: Clinical Institute Withdrawal Assessment for Alcohol Scale (CIWA-Ar) score ≥ 9; History of organic brain diseases or brain trauma; History of seizures, other neuropsychiatric disorders, or family history of psychiatric disorders; Presence of substance abuse/addiction other than alcohol (excluding nicotine addiction).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2024-06-30 (Estimated); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes in behavioral indicators of positive emotional attention bias towards alcohol-related cues | baseline, 1 day after treatment, 2 weeks after treatment
  Positive emotional attention bias is assessed through emotional attention bias under electroencephalogram recording, with the indicator being D scores calculated from the response time (D alcohol=RT (negative) - RT (positive) )/SD negative+positive).

SECONDARY OUTCOMES:
Changes in behavioral indicators of positive emotional attention bias towards healthy activity cues | baseline, 1 day after treatment, 2 weeks after treatment
  Positive emotional attention bias is assessed through emotional attention bias under electroencephalogram recording, with the indicator being D scores calculated from the response time (D health=RT (negative) - RT (positive) )/SD negative+positive).
Change of Craving assessed by Visual Analog Scale | baseline, 1 day after treatment, 2 weeks after treatment
  evaluate all participants' craving for for methamphetamine assessed by Visual Analog Scales (VAS). Score of VAS range from 0 to 10, and higher values represent high level of craving.
Change of Craving assessed by Visual Analog Mood Scale | baseline, 1 day after treatment, 2 weeks after treatment
  evaluate all participants' mood assessed by Visual Analog Scales (VAS). The scores ranges from 0 to 10, where 0 indicates the absence of the emotion and 10 indicates the emotion is extremely intense.

CONTACTS AND LOCATIONS:
Overall Officials: Min Zhao, Study Chair — Shanghai Mental Health Center

IPD SHARING:
Plan to Share IPD: No